CLINICAL TRIAL: NCT05485571
Title: Efficacy of Combined Microneedling With Methotrexate in Treatment of Alopecia Areata
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Asmaa Awad Hassanin, resident doctor at Dematology, Venereology and Andrology department at Gerga Hospital, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Soh-Med-22-07-07
Record Dates: First submitted 2022-07-24; First posted 2022-08-03 (Actual); Last update posted 2022-08-03 (Actual); Status verified 2022-08

CONDITIONS: Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GROUP 1 (Active Comparator): 15 patient with alopecia areata treated by microneedling only one session weekly for 12 weeks
  Interventions: Device: derma pen
- GROUP 2 (Active Comparator): 15 patient with alopecia areata treated by combined therapy with Microneedling and methotrexate After microneedling we applied methotrexate topically (25mg/ml) at dose 0.02ml/cm2 , A maximum of 0.1-0.2ml (2.5-5 mg) on the affected areas and rub it gently then Microneedling again, patient will take session weekly for 12 weeks.
  Interventions: Device: derma pen

INTERVENTIONS:
Device: derma pen — Group 1: Taking aseptic condition, 15 Patients were subjected to therapy with microneedling, patient will take session weekly for 12 weeks.
  Group 2: Taking aseptic condition, 15 patients were subjected to combined therapy with Microneedling and methotrexate After microneedling we applied methotrexate topically (25mg/ml) at dose 0.02ml/cm2 , A maximum of 0.1-0.2ml (2.5-5 mg) on the affected areas and rub it gently then Microneedling again, patient will take session weekly for 12 weeks
  Other Names: methotrexate

SUMMARY:
Alopecia areata (AA) is a common cause of non-cicatricial hair loss It is the second-most frequent non-scarring alopecia, after androgenic alopecia.

The prevalence of the disease is 0.2% in the general population with higher prevelance in younger (21-40 years of age) patients but no significant difference in incidence between males and females.

Several treatment options such as corticosteroids, anthralin, topical minoxidil, immunotherapy, and systemic therapy are commonly used with varying response . Unfortunately the traditional treatment options are frequently disappointing Available treatments may induce regrowth but do not modify the disease course .

Methotrexate (MTX) is a folic acid analog that binds to the dihydrofolate reductase enzyme, blocking the formation of tetrahydrofolate and so inhibits purine and pyrimidine metabolism and consequently nucleic acid synthesis. It acts as an immunosuppressant used in the treatment of several skin diseases Systemic MTX has been used in the treatment of AA, with satisfactory results. Microneedling is a minimally invasive procedure that utilizes multiple fine needles to create micropunctures in the skin.The act of creating these two to four cell-wide puncture holes triggers neovascularization, release of growth factors, and stimulates the expression of Wnt proteins. it has specifically been demonstrated to increase hair regrowth in alopecia via the release of platelet-derived growth factor, epidermal growth factors and activation of the hair bulge, all of which are triggered by the wound healing response .Increased expression of Wnt proteins, namely Wnt3a and Wnt10b, is also evident following microneedling. These particular proteins have been demonstrated to stimulate dermal papillae stem cells and hair growth.

ELIGIBILITY:
Inclusion Criteria:

- The study will include patients with alopecia areata

Exclusion Criteria:

* Children below 18 years , pregnant and lactating women .
* patients with chronic hepatic, hematological disorders or immunocompromised patients.
* patient recieved any treatment for alopecia areata in the last 3 months before the study.
* patients with extensive types (alopecia totalis, universalis and surface area >50%).

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-08-01 (Estimated); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
regrowth scale | 6 months
  0 score (regrowth < 10%) no response
  1. score (regrowth 11-25%) poor response
  2. score (regrowth 26-50%) fair response
  3. score (regrowth 51-75%) satisfactory response
  4. score (regrowth ≥ 75%) excellent response
Mcdonald Hull and Norris Regrowth Scale (by trichoscope) | 6 months
  Grade 1 - Regrowth of vellus hair. Grade 2 - Regrowth of sparse pigmented terminal hair. Grade 3 - Regrowth of terminal hair with patches of alopecia with patches of alopecia 50-75% in SALT score.
  Grade 4 - Regrowth of terminal hair on scalp with patches of alopecia > 75% in SALT score.

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag University Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Gilhar A, Paus R, Kalish RS. Lymphocytes, neuropeptides, and genes involved in alopecia areata. J Clin Invest. 2007 Aug;117(8):2019-27. doi: 10.1172/JCI31942. PMID 17671634
- [Background] Hou A, Cohen B, Haimovic A, Elbuluk N. Microneedling: A Comprehensive Review. Dermatol Surg. 2017 Mar;43(3):321-339. doi: 10.1097/DSS.0000000000000924. PMID 27755171
- [Background] Dhurat R, Sukesh M, Avhad G, Dandale A, Pal A, Pund P. A randomized evaluator blinded study of effect of microneedling in androgenetic alopecia: a pilot study. Int J Trichology. 2013 Jan;5(1):6-11. doi: 10.4103/0974-7753.114700. PMID 23960389
- [Background] Bressan AL, Silva RS, Fontenelle E, Gripp AC. [Immunosuppressive agents in Dermatology]. An Bras Dermatol. 2010 Jan-Feb;85(1):9-22. doi: 10.1590/s0365-05962010000100002. Portuguese. PMID 20464082